CLINICAL TRIAL: NCT05791370
Title: Red Palm Olein on Inflammation and Gut Health
Acronym: RPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: Universiti Putra Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PD232/18
Record Dates: First submitted 2022-12-20; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Diet; Healthy
Keywords: red palm olein; extra virgin coconut oil; extra virgin olive oil; high sensitivity C-reactive protein; inflammation; obesity
MeSH Terms: conditions — Inflammation; Obesity

STUDY DESIGN:
Intervention Model Description: We recruited a total of 156 overweight individuals, aged 25-45 years, with waist circumference ≥ 90 cm for men and ≥ 80 cm for women in a single-blind 3-arm randomised controlled trial. The participants consumed isocaloric diets (~ 2400 kcal) enriched with red palm olein (RPOO), extra virgin coconut oil (EVCO) and extra virgin olive oil (EVOO, as a control) for a 12-week duration
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: All data collected were blinded to the investigators by an independent third party until the completion of the analysis. The efficacy of the blinding procedure was assessed by evaluating the compliance of participants using the visual analogue scale to the experimental diets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Red palm olein (Experimental): Meals enriched with Red palm olein
  Interventions: Dietary Supplement: A 12-week parallel dietary intervention
- Extra virgin coconut oil (Experimental): Meals enriched with Extra virgin coconut oil
  Interventions: Dietary Supplement: A 12-week parallel dietary intervention
- Extra virgin olive oil (Experimental): Meals enriched with Extra virgin olive oil
  Interventions: Dietary Supplement: A 12-week parallel dietary intervention

INTERVENTIONS:
Dietary Supplement: A 12-week parallel dietary intervention — Subjects consumed 3 isocaloric meals prepared with the 3 oils for a duration of 12 weeks. The test meals were given for 5-day a week and contained 27-30% energy fat, with 2/3 (20% energy fat) replaced by experimental fat.

SUMMARY:
A parallel intervention was conducted to test the effect of consuming diets enriched with red palm olein (RPOO), extra virgin coconut oil (EVCO) and extra virgin olive oil (EVOO; positive control) in centrally obese individuals over a 12-week period. Following the screening of the subjects' health status, including their biochemical and lipid profiles, the subjects completed a 12-week dietary intervention. Both fasting blood and urine samples were collected at baseline (day 0) and endpoint (week 12); measurements were taken in duplicates. All data collected were blinded to the investigators by an independent third party until the completion of the analysis.

DETAILED DESCRIPTION:
The study was conducted according to the guidelines laid down in the Declaration of Helsinki. All subjects gave informed consent prior to the commencement of the study. A parallel intervention was conducted to test the effect of consuming diets enriched with red palm olein (RPOO), extra virgin coconut oil (EVCO) and extra virgin olive oil (EVOO; positive control) in centrally obese individuals over a 12-week period. Following the screening of the subjects' health status, including their biochemical and lipid profiles, the subjects completed a 12-week dietary intervention. Both fasting blood and urine samples were collected at baseline (day 0) and endpoint (week 12); measurements were taken in duplicates. All data collected were blinded to the investigators by an independent third party until the completion of the analysis. The efficacy of the blinding procedure was assessed by evaluating the compliance of participants using the visual analogue scale to the experimental diets. Statistical analysis was conducted independently by a statistician not involved in the conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

* aged 25-45 years
* waist circumference ≥ 90 cm for men and ≥ 80 cm for women

Exclusion Criteria:

* BMI ≤ 18.5 kg/m2
* medical history of cardiovascular diseases
* positive for diabetes or dyslipidemia
* diagnosed with chronic illness
* plasma total cholesterol > 6.5 mmol/L
* triacylglycerol >4.5 mmol/L
* on antihypertensive or lipid-lowering medication
* lactating
* pregnant
* smoking

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
hs-C reactive protein (hsCRP) | 12 weeks
  Changes in the mean of plasma hs-CRP at the endpoint relative to the baseline. Plasma hsCRP will be measured using an immunoturbidimetric method, fibrinogen by Clauss method (Dade)

SECONDARY OUTCOMES:
Plasma lipid profile: Total cholesterol (mmol/L) | 12 weeks
  Changes in the mean of plasma Total cholesterol (mmol/L) at the endpoint relative to the baseline. Total cholesterol analysis will be performed by enzymatic method by an accredited clinical laboratory (Pathology & Clinical Laboratory (M) Sdn. Bhd, Malaysia).
Plasma lipid profile: LDL cholesterol (mmol/L) | 12 weeks
  Changes in the mean of plasma LDL cholesterol (mmol/L) at the endpoint relative to the baseline. LDL cholesterol will be analysed by Friedewald calculation by an accredited clinical laboratory (Pathology & Clinical Laboratory (M) Sdn. Bhd, Malaysia).
Plasma lipid profile: HDL cholesterol (mmol/L) | 12 weeks
  Changes in the mean of plasma HDL cholesterol (mmol/L) at the endpoint relative to the baseline. Plasma HDL cholesterol will be analysed by elimination / catalase method by an accredited clinical laboratory (Pathology & Clinical Laboratory (M) Sdn. Bhd, Malaysia).
Plasma lipid profile: Triacylglycerol (mmol/L) | 12 weeks
  Changes in the mean of plasma Triacylglycerol (mmol/L) at the endpoint relative to the baseline. Plasma triglycerides will be analysed by glycerol phosphate oxidase method by an accredited clinical laboratory (Pathology & Clinical Laboratory (M) Sdn. Bhd, Malaysia).
Plasma lipid profile: Apolipoprotein B-100 (g/L) | 12 weeks
  Changes in the mean of plasma Apolipoprotein B-100 (g/L) at the endpoint relative to the baseline. Plasma apolipoprotein B-100 (apo B-100) will be analysed by PEG enhanced immunoturbidimetric method by an accredited clinical laboratory (Pathology & Clinical Laboratory (M) Sdn. Bhd, Malaysia).
Plasma lipid profile: Apolipoprotein A-1 (g/L) | 12 weeks
  Changes in the mean of plasma Apolipoprotein A-1 (g/L) at the endpoint relative to the baseline. Plasma Apolipoprotein A-1 will be analysed by PEG enhanced immunoturbidimetric method by an accredited clinical laboratory (Pathology & Clinical Laboratory (M) Sdn. Bhd, Malaysia).
Plasma fatty acid composition: Palmitic acid (C16:0) | 12 weeks
  Changes in the mean of plasma fatty acid composition (Palmitic acid (C16:0)) at the endpoint relative to the baseline. Lipids will be extracted from the plasma using Folch method and then trans-methylated with methanol and sulphuric acid. The fatty acid composition of the test fats will be determined by converting fatty acids of triacylglyceride to fatty acid methyl esters (FAME) according to AOCS Official Method Ch 1-91. The fatty acid composition will be determined according to AOCS Official Method Ce 1a-13 using Perkin Elmer Autosystem Gas Chromatography (PerkinElmer, Inc., California, USA). Data will be reported in g/100 g total fatty acids.
Plasma fatty acid composition: Oleic acid (C18:1 cis) | 12 weeks
  Changes in the mean of plasma fatty acid composition (Oleic acid (C18:1 cis)) at the endpoint relative to the baseline. Lipids will be extracted from the plasma using Folch method and then trans-methylated with methanol and sulphuric acid. The fatty acid composition of the test fats will be determined by converting fatty acids of triacylglyceride to fatty acid methyl esters (FAME) according to AOCS Official Method Ch 1-91. The fatty acid composition will be determined according to AOCS Official Method Ce 1a-13 using Perkin Elmer Autosystem Gas Chromatography (PerkinElmer, Inc., California, USA). Data will be reported in g/100 g total fatty acids.
Plasma fatty acid composition: Linoleic acid (C18:2n6 cis) | 12 weeks
  Changes in the mean of plasma fatty acid composition (Linoleic acid (C18:2n6 cis)) at the endpoint relative to the baseline. Lipids will be extracted from the plasma using Folch method and then trans-methylated with methanol and sulphuric acid. The fatty acid composition of the test fats will be determined by converting fatty acids of triacylglyceride to fatty acid methyl esters (FAME) according to AOCS Official Method Ch 1-91. The fatty acid composition will be determined according to AOCS Official Method Ce 1a-13 using Perkin Elmer Autosystem Gas Chromatography (PerkinElmer, Inc., California, USA). Data will be reported in g/100 g total fatty acids.
Plasma fatty acid composition: Linolenic acid (C18:3) | 12 weeks
  Changes in the mean of plasma fatty acid composition (Linolenic acid (C18:3)) at the endpoint relative to the baseline. Lipids will be extracted from the plasma using Folch method and then trans-methylated with methanol and sulphuric acid. The fatty acid composition of the test fats will be determined by converting fatty acids of triacylglyceride to fatty acid methyl esters (FAME) according to AOCS Official Method Ch 1-91. The fatty acid composition will be determined according to AOCS Official Method Ce 1a-13 using Perkin Elmer Autosystem Gas Chromatography (PerkinElmer, Inc., California, USA). Data will be reported in g/100 g total fatty acids.
Plasma antioxidant : alpha tocopherol (ug/ml) | 12 weeks
  Changes in the mean of plasma antioxidant (alpha tocopherol) at the endpoint relative to the baseline. The quantities of lipid-soluble antioxidants will be determined by reverse-phase HPLC (Agilent 1260 Infinity, US) and reported in ug/ml.
Plasma antioxidant : retinol (ug/ml) | 12 weeks
  Changes in the mean of plasma antioxidant (retinol) at the endpoint relative to the baseline. The quantities of lipid-soluble antioxidants will be determined by reverse-phase HPLC (Agilent 1260 Infinity, US) and reported in ug/ml.
Plasma antioxidant : alpha carotene (ug/ml) | 12 weeks
  Changes in the mean of plasma antioxidant (alpha carotene) at the endpoint relative to the baseline. The quantities of lipid-soluble antioxidants will be determined by reverse-phase HPLC (Agilent 1260 Infinity, US) and reported in ug/ml.
Plasma antioxidant : beta carotene (ug/ml) | 12 weeks
  Changes in the mean of plasma antioxidant (beta carotene) at the endpoint relative to the baseline. The quantities of lipid-soluble antioxidants will be determined by reverse-phase HPLC (Agilent 1260 Infinity, US) and reported in ug/ml.
Urinary Total Phenolics | 12 weeks
  Changes in the mean of urinary total phenolics at the endpoint relative to the baseline. Total phenolic content will be measured in urine samples using the Folin-Ciocalteu assay after a solid-phase clean-up
Dual-energy X-ray Absorptiometry (DEXA) Scan: Total body fat (z-score) | 12 weeks
  Changes in DEXA parameter (Total body fat (z-score)) at the endpoint relative to the baseline. DEXA scanning will be conducted in a subset of participants by trained personnel in the Prince Court Medical Centre, Malaysia with a Lunar Prodigy Advance densitometer (General Electric, Milwaukee, WI, USA).
Dual-energy X-ray Absorptiometry (DEXA) Scan: AP Spine (percentage of fat) | 12 weeks
  Changes in DEXA parameter (AP Spine (percentage of fat) at the endpoint relative to the baseline. DEXA scanning will be conducted in a subset of participants by trained personnel in the Prince Court Medical Centre, Malaysia with a Lunar Prodigy Advance densitometer (General Electric, Milwaukee, WI, USA).
Dual-energy X-ray Absorptiometry (DEXA) Scan: Left femur (percentage of fat) | 12 weeks
  Changes in DEXA parameter (Total body fat (Left femur (percentage of fat) at the endpoint relative to the baseline. DEXA scanning will be conducted in a subset of participants by trained personnel in the Prince Court Medical Centre, Malaysia with a Lunar Prodigy Advance densitometer (General Electric, Milwaukee, WI, USA).
Dual-energy X-ray Absorptiometry (DEXA) Scan: BMD AP spine L1-L4 (g/cm2) | 12 weeks
  Changes in DEXA parameter (BMD AP spine L1-L4 (g/cm2)) at the endpoint relative to the baseline. DEXA scanning will be conducted in a subset of participants by trained personnel in the Prince Court Medical Centre, Malaysia with a Lunar Prodigy Advance densitometer (General Electric, Milwaukee, WI, USA).
Dual-energy X-ray Absorptiometry (DEXA) Scan: AP spine L1-L4 (z-score) | 12 weeks
  Changes in DEXA parameter (AP spine L1-L4 (z-score)) at the endpoint relative to the baseline. DEXA scanning will be conducted in a subset of participants by trained personnel in the Prince Court Medical Centre, Malaysia with a Lunar Prodigy Advance densitometer (General Electric, Milwaukee, WI, USA).
Dual-energy X-ray Absorptiometry (DEXA) Scan: BMD total femur (g/cm2) | 12 weeks
  Changes in DEXA parameter (BMD total femur (g/cm2)) at the endpoint relative to the baseline. DEXA scanning will be conducted in a subset of participants by trained personnel in the Prince Court Medical Centre, Malaysia with a Lunar Prodigy Advance densitometer (General Electric, Milwaukee, WI, USA).
Gut Microbiome: Alpha and Beta Diversities | 12 weeks
  Changes in gut microbiome data: Alpha and Beta Diversities at the endpoint relative to the baseline. The analyses will be done on the complete OTU count table. Sample ordination in principal coordinate axis (PCoA) space will be visualised using the first two principal coordinate axes. NGS Amplicon sequencing and gut microbiota analyses will be performed by Apical Scientific Sdn Bhd.
Gut Microbiome: Firmicutes to Bacteroides Ratio | 12 weeks
  Changes in gut microbiome (Firmicutes to Bacteroides Ratio) at the endpoint relative to the baseline. Computation of Firmicutes to Bacteroides (F/B) ratio using the complete microbial count table. NGS Amplicon sequencing and gut microbiota analyses will be performed by Apical Scientific Sdn Bhd.
Gut Microbiome: Differential Abundance Analysis | 12 weeks
  Changes in gut microbiome (Differential Abundance Analysis) at the endpoint relative to the baseline. NGS Amplicon sequencing and gut microbiota analyses will be performed by Apical Scientific Sdn Bhd.
Plasma inflammatory marker: IL-6 (pg/mL) | 12 weeks
  Changes in Plasma inflammatory marker: IL-6 (pg/mL) at the endpoint relative to the baseline. Plasma IL-6 will be measured by quantitative sandwich enzyme immunoassay (R&D Systems, USA).
Plasma inflammatory marker: IL-1beta (pg/mL) | 12 weeks
  Changes in Plasma inflammatory marker:IL-1beta (pg/mL) at the endpoint relative to the baseline. Plasma IL-1beta will be measured by quantitative sandwich enzyme immunoassay (R&D Systems, USA).
Plasma inflammatory marker: TNF-alpha (pg/mL) | 12 weeks
  Changes in Plasma inflammatory marker: TNF-alpha (pg/mL) at the endpoint relative to the baseline. Plasma TNF-alpha will be measured by quantitative sandwich enzyme immunoassay (R&D Systems, USA).
Plasma inflammatory marker: sICAMs (ng/mL) | 12 weeks
  Changes in Plasma inflammatory marker: sICAMs (ng/mL) at the endpoint relative to the baseline. Plasma sICAM-1 will be measured by quantitative sandwich enzyme immunoassay (R&D Systems, USA).
Plasma inflammatory marker: sVCAMs (ng/mL) | 12 weeks
  Changes in Plasma inflammatory marker: sVCAMs (ng/mL) at the endpoint relative to the baseline. Plasma sVCAM-1 will be measured by quantitative sandwich enzyme immunoassay (R&D Systems, USA).
Plasma inflammatory marker: RBP-4 (ng/mL) | 12 weeks
  Changes in Plasma inflammatory marker: RBP4 at the endpoint relative to the baseline. Plasma RBP-4 will be measured by quantitative sandwich enzyme immunoassay (R&D Systems, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Kim Tiu Teng, PhD, Principal Investigator — Malaysia Palm Oil Board
Locations (1):
- Malaysian Palm Oil Board, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the individual participant data , provided requested specifically for scientific analysis purposes

REFERENCES:
- [Derived] Teng KT, Loganathan R, Chew BH, Khang TF. Diverse impacts of red palm olein, extra virgin coconut oil and extra virgin olive oil on cardiometabolic risk markers in individuals with central obesity: a randomised trial. Eur J Nutr. 2024 Jun;63(4):1225-1239. doi: 10.1007/s00394-024-03338-6. Epub 2024 Feb 19. PMID 38372798